CLINICAL TRIAL: NCT05679960
Title: Point of Care, Real-Time Urine Metabolomics Test to Diagnose Colorectal Cancers and Polyps in Low-and Middle-Income Countries
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The urine POC device seems not to be promising in colorectal cancer screening
Sponsor: Obafemi Awolowo University Teaching Hospital (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); University of Alberta (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Olusegun Alatise, Professor/Consultant Surgeon, Obafemi Awolowo University Teaching Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NHREC/01/01/2007-18/10/2021
Record Dates: First submitted 2022-07-26; First posted 2023-01-11 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients low gastrointestinal tract bleeding (Active Comparator): Patients presenting in the surgical outpatients or emergency department with low gastrointestinal tract bleeding
  Interventions: Diagnostic Test: Urine PolypDx machine Versus Colonoscopy
- Participants who are high risk due to a family history of CRC (Active Comparator): First degree relatives of patients diagnosed with colorectal cancer
  Interventions: Diagnostic Test: Urine PolypDx machine Versus Colonoscopy
- Patients with a diagnosis of stage I-III CRC who have no evidence of disease (Active Comparator): Patients previously diagnosed of stage I-III CRC and managed in the hospital but are now having no evidence of disease
  Interventions: Diagnostic Test: Urine PolypDx machine Versus Colonoscopy

INTERVENTIONS:
Diagnostic Test: Urine PolypDx machine Versus Colonoscopy — 1. Urine samples of the participants in each group will be analyzed to check for preidentified metabolites that signified colorectal cancer
  2. Colonoscopy, which is the gold standard for colorectal cancer diagnosis/screening will be performed on all the participants positive for metabolites signifying CRC on Urine PolypDx machine in all the groups

SUMMARY:
Study description: the study is a clinical trial aimed at assessing the validity of a point-of-care tool developed for colorectal cancer screening using urine metabolites.

Objectives:

Primary Objective:

In the pilot phase, investigators will field test the POC device in Nigeria on 75 patients who are high-risk for CRC and then validate the urine metabolite signature using a large cohort of 645 patients at high risk for CRC and polyps. This will allow us to determine the sensitivity and specificity of this device and these signatures for CRC and polyps.

Endpoints: the endpoint will be the calculation of the validity (sensitivity and specificity) of the tool. Positive and negative predictive values will also be calculated.

Study population:

Patients > 40 years of age with LGI bleeding for more than one-week OR

* Patients who are high risk due to a family history of CRC (first-degree relative)
* Must be at most 10 years younger than when relative presented with CRC (For example, a patient with a relative diagnosed at age 40 with CRC will be eligible after age 30)
* Patients with a diagnosis of stage I-III CRC who have no evidence of disease Both males and females will be involved in the study

I. The study will evaluate the validity and acceptability of the POC biosensor device in Nigeria.

Description of sites/facilities enrolling participants: the study will be conducted at Obafemi Awolowo University Teaching Hospitals Complex (OAUTHC) which hosts the head office of African Research Group for Oncology (ARGO). The study will also run concurrently at other ARGO collaborating sites. All the ARGO collaborating sites are tertiary health care facilities with experienced personnel to oversee the study. The pilot study will, however, take place in OAUTHC alone.

Study duration:

The accrual time for the validation study is 2.5 years. Participant Duration: the study will require initial one-time contact. Those that are positive during the screening with the POC biosensor device will be booked for colonoscopy. Hence, for participants with positive results to complete the study may require 2 weeks on average.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 40 years of age with LGI bleeding for more than one week OR
* Patients who are high risk due to a family history of CRC (first-degree relative)
* Must be at most 10 years younger than when relative presented with CRC (For example, a patient with a relative diagnosed at age 40 with CRC will be eligible after age 30)
* Patients with a diagnosis of stage I-III CRC who have no evidence of disease

Exclusion Criteria:

criteria

* Patients who are unable to provide written informed consent;
* Previous diagnosis, treatment, or surgery for any cancer other than CRC
* Age younger than 40 years with no family history of CRC
* Any significant medical comorbidities that the anesthesiologist or surgeon determines is a contraindication for colonoscopy in their facility.
* Inability to provide a urine sample no fewer than 3 days before colonoscopy.
* Inability to fully complete the patient satisfaction survey tool
* Diagnosis of or suspected inflammatory bowel disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 645 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Urine PolypDx device in detecting colorectal cancer | One month
  Results from the urine assay will be compared with the histology report of the tissue taken during colonoscopy, the gold standard for colorectal cancer diagnosis. Sensitivity, specificity, positive predictive value, and negative predictive values will be calculated

SECONDARY OUTCOMES:
Sensitivity Urine PolypDx device in detecting colorectal cancer (CRC) | One month
  Proportion of those urine PolyDx device detects to have CRC that actually have CRC
Specificity Urine PolypDx device in detecting colorectal cancer (CRC) | One month
  Proportion of those urine PolyDx device detects not to have CRC that actually do not have CRC
Positive Predictive Value Urine PolypDx device in detecting colorectal cancer (CRC) | One month
  Proportion of those who test positive with urine PolyDx device that actually do have CRC that actually have CRC
Negative Predictive Value Urine PolypDx device in detecting colorectal cancer (CRC) | One month
  Proportion of those who test negative with urine PolyDx device that actually do not have CRC that actually have CRC

CONTACTS AND LOCATIONS:
Locations (1):
- Obafemi Awolowo University Teaching Hospital, Ile-Ife, Osun State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available after publication of the data
Access Criteria: Data will be made accessible upon reasonable request directed to the principal investigator of this study by any researcher in related fields